CLINICAL TRIAL: NCT01335906
Title: A Randomized Trial of an Evidence-informed Choice Based on Appreciation of Risks and Benefits for Women Participating in Mammography Screening
Brief Title: Evidence-informed Choice for Women Participating in Mammography Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, José Manuel Baena Cañada, MD, PhD, Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: PI-0315-2010
Record Dates: First submitted 2011-04-06; First posted 2011-04-15 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Early Detection of Cancer
Keywords: Cancer Screening Tests; Early Diagnosis of Cancer; Mammography; Informed Consent; Consent Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evidence-based informed consent (Experimental)
  Interventions: Other: Information
- Usual information (No Intervention)

INTERVENTIONS:
Other: Information — The experimental information consists of receiving verbal and written evidence-based information about the benefits and risks of mammography screening program. The standard information consists of receiving the information that public institutions provide to the women invited to the screening program.
  Arms: Evidence-based informed consent

SUMMARY:
Study objectives: to evaluate the effects of information about benefits and risks of mammography screening on participants in terms of knowledge, attitude, rates of uptake, fear of cancer, anxiety, and conflict decision. Study hypothesis: information about benefit and risks of mammography screening increases the women´s knowledge of it; allows women to make an informed decision on whether to stop or continue the screening program, changing the actual participation rate; anxiety and fear are not increased. Design: randomized controlled clinical trial with non-pharmacological intervention. Subjects and setting of study: women referred to mammography screening in the District Bay of Cádiz-La Janda. Interventions: random assignment of women in two arms according to the information provided. Control arm is the standard information; it consists of receiving information normally provided to women attending the screening program for breast cancer. Intervention arm is the experimental information and consists of receiving accurate verbal and written information about the benefits and real risks of mammography screening programs by a physician investigator. Determinations: knowledge, attitude, rates of uptake, fear of cancer, anxiety, and conflict decision.

ELIGIBILITY:
Inclusion Criteria:

* Women living in the Bay Health District Cádiz-La Janda
* Women aged between 45 and 69 years
* Women invited to breast screening program and who attend it
* Qualified women to give informed consent to participate in the study

Exclusion Criteria:

* Women with a history of breast cancer

Ages: 45 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knowledge of women participating in the screening program | Before randomization (baseline) and one month later
  The primary outcome measure is the level of knowledge obtained in a specific questionnaire, in which there are 7 questions, of which 3 are quantitative with no assumptions and are scored with 2 points. There are also 4 qualitative questions that have 3 assumptions which are scored with 1 point. The maximum score is 10 and minimum 0. It is considered that a woman has made a choice based on adequate knowledge if she gets a score of 6 or more.

SECONDARY OUTCOMES:
Attitudes, intention to participate, fear and anxiety of women participating in the screening program | Before randomization (baseline) and one month later. Two years later, women will be called to the follow-up mammography. At this time the real choice taken by woman will be investigated
  The investigators will investigate whether the attitudes of women towards mammography screening are positive or negative. They will respond to 4 questions that are scored from 0 to 6. To know their decision whether to participate in mammography screening they will answer "I am determined to participate" "I am determined not to participate" and "I am undecided". Effective participation will be investigated 2 years later. The level of anxiety and fear of cancer will be measured by "Hospital Anxiety and depression" scale.

CONTACTS AND LOCATIONS:
Overall Officials: José M Baena-Cañada, MD, PhD, Study Chair — Oncology Unit, University Hospital Puerta del Mar, Cádiz; Petra Rosado, MD, Study Director — Oncology Unit, University Hospital Puerta del Mar, Cádiz; Inmaculada Expósito, Chemistry, Principal Investigator — Oncology Unit, University Hospital Puerta del Mar, Cádiz; María del Carmen Díaz, Chemistry, Principal Investigator — Oncology Unit, University Hospital Puerta del Mar, Cádiz; Juan Nieto, MD, Principal Investigator — Health District Bay of Cádiz-La Janda
Locations (1):
- Oncology Unit, Puerta del Mar University Hospital, Cadiz, Andalusia, Spain